CLINICAL TRIAL: NCT01023672
Title: An Open Label, Single-Center Pilot Study of Armodafinil in Patients With Dementia With Lewy Bodies
Brief Title: "Pilot Study of Armodafinil in Patients With Dementia With Lewy Bodies"
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Cephalon (Industry); National Institute on Aging (NIA) (NIH)
Responsible Party: Bradley F. Boeve, MD, Mayo Clinic Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-003438; R01AG015866 (NIH); P50AG016574 (NIH)
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Results first posted 2013-09-05 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-06

CONDITIONS: Dementia With Lewy Bodies
Keywords: Dementia with Lewy Bodies; hypersomnolence; cognition; neuropsychiatric morbidity; quality of life
MeSH Terms: conditions — Lewy Body Disease; Disorders of Excessive Somnolence | interventions — Modafinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Armodifinil (Other): 150-250 mg armodafinil by mouth daily
  Interventions: Drug: Armodafinil

INTERVENTIONS:
Drug: Armodafinil — 150-250 mg armodafinil by mouth daily
  Other Names: Nuvigil

SUMMARY:
This research study is to examine the effects of the study medication Armodafinil in patients with dementia with Lewy bodies (DLB).

DLB is associated with memory and other thinking problems, excessive daytime sleepiness, hallucinations, delusions, apathy, and reduced quality of life.

One type of medication that could potentially improve daytime sleepiness, memory and thinking skills, hallucinations, delusions, apathy, and quality of life is known as a wake-promoting medication. Armodafinil is a wake-promoting medication that has been developed for treatment of patients with narcolepsy, sleep apnea, and other disorders which cause excessive daytime sleepiness.

The drug used in this study is considered investigational, which means it has either not been approved by the Food and Drug Administration (FDA) for routine clinical use or for the use described in this study. However the FDA has allowed the use of this drug/device in this research study.

In this study, patients with DLB will receive daily oral Armodafinil tablets, and their response to treatment will be assessed over 12 weeks. This study does not involve any placebo medication, so all patients will receive Armodafinil treatment.

DETAILED DESCRIPTION:
In patients with DLB, the following aims/objectives will be addressed by comparing data on key measures at baseline and at 4 and 12 weeks of therapy:

Primary Aims - to test the hypotheses that armodafinil therapy at 150-250 mg every morning:

* will result in improvement in excessive daytime sleepiness as measured by the Epworth Sleepiness Scale (ESS) and Maintenance of Wakefulness Test (MWT) (Aim 1A)
* will result in improvement in the cognitive subscale of the Alzheimer's Disease Assessment Scale (ADAS-Cog) (Aim 1B)
* will result in improvement in the Alzheimer's Disease Cooperative Study-Clinician's Global Impression of Change (ADCS-CGIC) (Aim 1C)
* will be well-tolerated with no significant side-effects present (Aim 1D)

Secondary Aims - to test the hypotheses that armodafinil therapy at 150-250 mg every morning will result in improvement in:

* cognition as measured by the Mini-Mental State Examination (MMSE) and other focused neuropsychological tests (Aim 2A)
* neuropsychiatric morbidity, particularly apathy, depression, visual hallucinations, and delusions, as measured by the Neuropsychiatric Inventory (NPI) (Aim 2B)
* functional status as measured by the Alzheimer's Disease Cooperative Study-Activities of Daily Living (ADCS-ADL) (Aim 2C)
* patient and caregiver quality of life (QOL) as measured by the linear analog scale (LASA) (Aim 2D)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of clinically possible or probable DLB using established criteria
* Age 50-90 inclusive
* Epworth Sleepiness Scale score of 8 or greater
* MMSE score between 10 and 26 inclusive
* No active medical disorder that could preclude participation in a drug treatment trial over a 12 week protocol
* Stable medication regimen over previous four weeks
* Absence of psychotropic medications at doses viewed by the clinician to be significantly impacting the patient's alertness during wakefulness
* Absence of clinically significant primary sleep-related breathing disorder causing sleepiness as demonstrated by polysomnography (PSG) [ie, no significant upper airway resistance syndrome (UARS), obstructive sleep apnea (OSA), nor central sleep apnea (CSA) as reflected by a combined respiratory disturbance index (RDI) <15] OR adequate documentation of efficacy of treatment for UARS, OSA, and CSA
* Caregiver that is with the patient at least 4 hours/day for at least 5 days per week
* Patient and caregiver willing and able to participate in all study-related procedures
* Patient is capable of giving informed consent, or if appropriate, has caregiver capable of giving consent on the subject's behalf.

Exclusion Criteria:

* Does not fulfill criteria for clinically possible or probable DLB
* Age <50 or >90
* Women with intact uterus and not post-menopausal unless pregnancy test performed at screening is negative
* Epworth Sleepiness Scale score less than 8
* MMSE score <10 or >26
* Active medical disorder that could preclude participation in a drug treatment trial over a 52 week protocol, such as:

  * Hypertension with BP readings exceeding 150 mm Hg systolic and 90 mm Hg diastolic
  * Hypersensitivity to modafinil, armodafinil, or any other conventional stimulants
  * Myocardial infarction or cerebral infarct over preceding year, stable or unstable angina, known symptomatic coronary artery disease
  * History of left ventricular hypertrophy or mitral valve prolapse
  * History of chronic or paroxysmal atrial fibrillation, chronic or paroxysmal atrial flutter, ventricular fibrillation, or ventricular tachycardia
  * History of cancer over preceding 1 year (excluding squamous or basal cell carcinoma of the skin)
  * History of Stevens-Johnson syndrome (SJS), toxic epidermal necrolysis (TEN), and drug rash with eosinophilia and systemic symptoms (DRESS)
  * Pulmonary disease requiring oral or inhalatory medications
  * Any other medical disorder considered by the study physicians as inappropriate for any wake-promoting medication
* Medication regimen has not been stable over preceding four weeks
* Concurrent use of lamotrigine or oxcarbazepine
* Presence of over-the-counter and prescription psychotropic medications at doses viewed by the clinician to be significantly impacting the patient's alertness during wakefulness, such as:

  * Clonazepam > 1 mg/night
  * Seroquel > 100 mg/night
  * Zyprexa > 10 mg/night
* Presence of another clinically-significant primary sleep disorder (eg, UARS, OSA, CSA) that is not being treated
* Clinically significant abnormalities on screening ECG or laboratory tests
* Patient or caregiver unwilling or unable to participate in all study-related procedures
* Caregiver is not with patient at least 4 hours/day for at least 5 days/week
* Patient or caregiver unwilling or unable to provide informed consent
* CT or MRI evidence of a clinically significant structural lesion that could account for the participants dementia

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley F Boeve, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at the Mayo Clinic in Rochester, Minnesota
Period: Overall Study
Arm/Group | Armodifinil
Started | 20
Completed | 17
Not Completed | 3
Not completed — Worsening disease | 2
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Armodifinil
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Mean Initial Sleep Latency as Measured by the Maintenance of Wakefulness Test (MWT)
Description: The MWT measures the subject's ability to stay awake while sitting quietly in a chair. The test has 4 parts, each lasting 40 minutes if the subject is able to remain awake that long each time, and the parts are spaced apart in 2 hour intervals through the day.
  The subject is placed in a dim room, with the only source of light slightly behind the subject's head and out of his/her field of vision, and back and neck supported. During this time the subject is monitored with the same measures that are used in a standard overnight sleep study called a polysomnogram. The sleep latency, or time it takes the subject to fall asleep, will be recorded.
  In healthy people, the time it takes to fall asleep may be approximately 30 minutes on the test. More than 97% of people will take eight minutes or longer to fall asleep. Therefore, sleep latency that is less than eight minutes is considered to be abnormal.
Time Frame: baseline, 12 weeks
Population: Per Protocol; 3 subjects did not complete the study (2 had worsening disease, and 1 died) and did not complete this test.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Armodifinil
Number analyzed (Participants) | 17
minutes
  Baseline | 7.0 [4.25 to 19.07]
  12 Weeks | 19.0 [7.19 to 32.76]
Statistical Analysis 1: Comparison: Armodifinil; The analysis was done per protocol (n=17); Test type: Superiority or Other; p = 0.003, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Subjects were followed for adverse events from the initiation of any study procedure until 30 days following the last administration of study treatment.
Arm/Group | Armodifinil
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 5/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Armodifinil (N=20)
Anxiety (Psychiatric disorders) | 1 (2)
Blepharitis (Eye disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
ECG changes/prolonged QTc interval (Cardiac disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Otalgia (Ear and labyrinth disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No